CLINICAL TRIAL: NCT02301975
Title: A Randomized, Double-blind, Double-dummy, Parallel Group, Multicenter Study of Once Daily Fluticasone Furoate/Vilanterol 100/25 mcg Inhalation Powder, Twice Daily Fluticasone Propionate/Salmeterol 250/50 mcg Inhalation Powder, and Twice Daily Fluticasone Propionate 250 mcg Inhalation Powder in the Treatment of Persistent Asthma in Adults and Adolescents Already Adequately Controlled on Twice-daily Inhaled Corticosteroid and Long-acting beta2 Agonist
Brief Title: An Efficacy and Safety Study of Fluticasone Furoate/Vilanterol 100/25 Microgram (mcg) Inhalation Powder, Fluticasone Propionate/Salmeterol 250/50 mcg Inhalation Powder, and Fluticasone Propionate 250 mcg Inhalation Powder in Adults and Adolescents With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201378
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: Adult; asthma; Fluticasone Propionate; Adolescents; Salmeterol; Vilanterol; ELLIPTA; ACCUHALER/DISKUS; Non-inferior; Fluticasone Furoate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone Furoate/Vilanterol 100/25 mcg (Experimental): FF/VI 100/25 mcg by inhalation OD (PM) via ELLIPTA plus placebo by inhalation BD (AM and PM) via ACCUHALER/DISKUS for 24 weeks.
  Interventions: Drug: Fluticasone Furoate/Vilanterol 100/25 mcg via ELLIPTA inhaler; Drug: Placebo inhalation powder via ACCUHALER/DISKUS inhaler
- Fluticasone Propionate/Salmeterol 250/50 mcg (Experimental): FP/Salmeterol 250/50 mcg by inhalation BD (AM and PM) via ACCUHALER/DISKUS plus placebo by inhalation OD (PM) via ELLIPTA for 24 weeks.
  Interventions: Drug: Placebo inhalation powders via ELLIPTA inhaler; Drug: Fluticasone Propionate/Salmeterol 250/50 mcg via ACCUHALER/DISKUS inhaler
- Fluticasone Propionate 250 mcg (Experimental): FP 250 mcg by inhalation BD (AM and PM) via ACCUHALER/DISKUS plus placebo by inhalation OD (PM) via ELLIPTA for 24 weeks.
  Interventions: Drug: Placebo inhalation powders via ELLIPTA inhaler; Drug: Fluticasone Propionate 250 mcg via ACCUHALER/DISKUS inhaler

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol 100/25 mcg via ELLIPTA inhaler — FF/Vilanterol 100/25 mcg inhalation powders administered once daily via ELLIPTA inhaler. 30 doses per device and 100/25 mcg per actuation.
  Arms: Fluticasone Furoate/Vilanterol 100/25 mcg
Drug: Placebo inhalation powders via ELLIPTA inhaler — Placebo inhalation powders administered once daily via ELLIPTA inhaler. 30 doses per device.
  Arms: Fluticasone Propionate 250 mcg; Fluticasone Propionate/Salmeterol 250/50 mcg
Drug: Fluticasone Propionate/Salmeterol 250/50 mcg via ACCUHALER/DISKUS inhaler — FP/Salmeterol 250/50 mcg inhalation powder administered twice daily via ACCUHALER/DISKUS inhaler. 60 doses per device and 250/50 mcg per actuation.
  Arms: Fluticasone Propionate/Salmeterol 250/50 mcg
Drug: Placebo inhalation powder via ACCUHALER/DISKUS inhaler — Placebo inhalation powder administered twice daily via ACCUHALER/DISKUS inhaler. 60 doses per device.
  Arms: Fluticasone Furoate/Vilanterol 100/25 mcg
Drug: Fluticasone Propionate 250 mcg via ACCUHALER/DISKUS inhaler — FP 250 mcg inhalation powder administered twice daily via ACCUHALER/DISKUS inhaler. 60 doses per device and 250 mcg per actuation.
  Arms: Fluticasone Propionate 250 mcg

SUMMARY:
This study is a randomized, double-blind, double-dummy, parallel group, multicenter, non-inferiority study. The study will enroll adult and adolescent asthmatic subjects who are currently receiving mid dose inhaled corticosteroids (ICS) plus long-acting beta2-agonist (LABA) (equivalent to fluticasone propionate [FP]/salmeterol 250/50 microgram [mcg]twice daily [BD]), either via a fixed dose combination product or through separate inhalers. The study consists of a LABA washout period of 5 days and a run-in period of 4 weeks, followed by a treatment period of 24 weeks, and a follow up contact period of one week. The total duration of the study is 30 weeks. Approximately 1461 subjects will be randomized to one of the following three treatments (487 per treatment): fluticasone furoate (FF)/vilanterol (VI) 100/25 mcg once daily (OD) in the evening (PM) via ELLIPTA™ inhaler plus placebo BD via ACCUHALER™/DISKUS™; FP/salmeterol 250/50 mcg BD via ACCUHALER/DISKUS inhaler plus placebo OD (PM) via ELLIPTA inhaler; FP 250 mcg BD via ACCUHALER/DISKUS inhaler plus placebo OD (PM) via ELLIPTA inhaler. In addition, all subjects will be supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms. This study will determine if FF/VI 100/25 mcg OD via ELLIPTA inhaler is non-inferior to FP/salmeterol 250/50 mcg BD via ACCUHALER/DISKUS inhaler in adult and adolescent asthmatic subjects already adequately controlled on a twice-daily ICS/LABA.

SERETIDE, ELLIPTA, ACCUHALER, RELVAR, and DISKUS are trademarks of the GlaxoSmithKline Group of Companies.

ELIGIBILITY:
Inclusion Criteria

* Subjects must give their signed and dated written informed consent to participate prior to commencing any study related activities.
* Subjects must be outpatients >=12 years of age at Visit 1 who have had a diagnosis of asthma, as defined by the National Institutes of Health, for at least 12 weeks prior to Visit 1 (Note: Countries with local restrictions prohibiting enrollment of adolescents will enroll subjects >=18 years of age only).
* Subjects may be male or an eligible female. An eligible female is defined as having non-childbearing potential or having childbearing potential and a negative urine pregnancy test at Screening and agrees to use an acceptable method of birth control consistently and correctly.
* Subjects must have a FEV1 of >=80% of the predicted normal value.
* Subjects are eligible if they have received mid dose ICS plus LABA (equivalent to FP/salmeterol 250/50 twice daily or an equivalent combination via separate inhalers) for at least the 12 weeks immediately preceding Visit 1.
* All subjects must be able to replace their current SABA treatment with albuterol/salbutamol aerosol inhaler at Visit 1 for use, as needed, for the duration of the study. Subjects must be able to withhold albuterol/salbutamol for at least 6 hours prior to study visits.
* If in the opinion of the investigator the subject's asthma is well controlled. Exclusion Criteria
* History of Life-Threatening Asthma, defined for this protocol as an asthma episode that required intubation and/or associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 5 years.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or in the opinion of the Investigator, expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Any asthma exacerbation requiring oral corticosteroids within 12 weeks of Visit 1 or resulting in an overnight hospitalization requiring additional treatment for asthma within 6 months prior to Visit 1.
* A subject must not have current evidence of Atlectasis, Bronchopulmonary dysplasia, Chronic bronchitis, Chronic obstructive pulmonary disease, Pneumonia, Pneumothorax, Interstitial lung disease, or any evidence of concurrent respiratory disease other than asthma
* A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study.
* A subject must not have used any investigational drug within 30 days prior to Visit 1 or within five half-lives (t½) of the prior investigational study, whichever is longer of the two.
* Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of RELVAR™ ELLIPTA inhaler, SERETIDE™ ACCUHALER/DISKUS inhaler or FP 250.
* History of severe milk protein allergy.
* Administration of prescription or non-prescription medication that would significantly affect the course of asthma, or interact with study drug.
* A subject must not be using or require the use of immunosuppressive medications during the study.
* A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location which seems likely (in the opinion of the Investigator) to impair compliance with any aspect of this study protocol, including visit schedule and completion of the daily diaries.
* Current tobacco smoker or has a smoking history of 10 pack-years (20 cigarettes/day for 10 years). A subject may not have used inhaled tobacco products or inhaled marijuana within the past 3 months (e.g., cigarettes, cigars, electronic cigarettes, or pipe tobacco).
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1526 (Actual)
Dates: Start 2015-03-01; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (142):
- United States (33):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Hendersonville, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Greenfield, Wisconsin
- Argentina (9):
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Brazil (4):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo
- Chile (5):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Viña del Mar
- Czechia (11):
  - GSK Investigational Site, Česká Lípa
  - GSK Investigational Site, Hlučín
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Kutná Hora
  - GSK Investigational Site, Lovosice
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Varnsdorf
- Germany (23):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Peine, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Mexico (5):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mexico City
- Netherlands (9):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Zutphen
- Romania (10):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (19):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Vladimir
  - GSK Investigational Site, Volgodonsk
  - GSK Investigational Site, Voronezh
- South Korea (4):
  - GSK Investigational Site, Cheongju-si, Chungcheongbuk-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
- Spain (10):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Bernstein D, Andersen L, Forth R, Jacques L, Yates L. Once-daily fluticasone furoate/vilanterol versus twice-daily fluticasone propionate/salmeterol in patients with asthma well controlled on ICS/LABA. J Asthma. 2018 Sep;55(9):984-993. doi: 10.1080/02770903.2017.1386214. Epub 2018 Apr 13. PMID 28961020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants at screening and run-in visits entered a 24 Week treatment period and were randomized to receive either Fluticasone furoate/Vilanterol (FF/VI) 100/25 micrograms (mcg) or Fluticasone propionate/salmeterol (FP/S) 250/50mcg or only FP 250mcg followed by a follow-up phase. The total duration for study participation was 30 weeks.
Pre-assignment Details: A total of 3162 adult and adolescent participants with asthma were screened, out of which 516 were screen-failures, 1124 were run-in failures, 1522 participants were randomized, and 1504 subjects received at least one dose of study medication to be included in the Intent-to-Treat (ITT) Population.
Groups:
- FF/VI 100/25 mcg Once Daily: Participants received FF/VI 100/25 mcg via ELLIPTA® inhaler once daily (at evening) along with placebo via ACCUHALER/DISKUS® twice daily for 24 weeks. Albuterol/Salbutamol inhalation aerosol was also provided to treat acute asthma symptoms.
- FP/S 250/50 mcg Twice Daily: Participants received FP/S 250/50 mcg via ACCUHALER/DISKUS inhaler twice daily along with placebo via ELLIPTA inhaler once daily (at evening) for 24 weeks. Albuterol/Salbutamol inhalation aerosol was also provided to treat acute asthma symptoms.
- FP 250 mcg Twice Daily: Participants received FP 250 mcg via ACCUHALER/DISKUS inhaler twice daily along with placebo via ELLIPTA inhaler once daily (at evening) for 24 weeks. Albuterol/Salbutamol inhalation aerosol was also provided to treat acute asthma symptoms.
Period: Overall Study
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Started | 504 | 501 | 499
Completed | 473 | 476 | 477
Not Completed | 31 | 25 | 22
Not completed — Adverse Event | 8 | 3 | 2
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Protocol Violation | 3 | 5 | 3
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Physician Decision | 4 | 2 | 3
Not completed — Withdrawal by Subject | 15 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily | Total
Number analyzed (Participants) | 504 | 501 | 499 | 1504
Age, Continuous [Mean (Standard Deviation); unit: Participants] | 44.4 (16.30) | 43.0 (15.20) | 43.0 (16.58) | 43.5 (16.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 336 | 314 | 964
  Male | 190 | 165 | 185 | 540
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska native | 0 | 0 | 1 | 1
  Asian - East Asian Heritage | 8 | 11 | 4 | 23
  Asian- Japanese Heritage | 1 | 0 | 0 | 1
  Asian- South East Asian Heritage | 1 | 0 | 1 | 2
  Black/African American Heritage | 12 | 14 | 17 | 43
  White- Arabic/ North African Heritage | 0 | 1 | 2 | 3
  White- White/Caucasian/European Heritage | 415 | 407 | 410 | 1232
  White- Mixed White Race | 1 | 0 | 0 | 1
  African American/ African and White Heritage | 0 | 5 | 0 | 5
  American Indian/Alaskan Native and White Heritage | 66 | 62 | 64 | 192
  Asian - East Asian and White Heritage | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Evening (Post Meridiem [PM]) Forced Expiratory Volume in One Second (FEV1) Using Intent-to-Treat (ITT) Population
Description: FEV1 was defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 (pre-bronchodilator and pre-dose) was measured at Baseline up to Week 24 at evening using spirometry. Repeated Measures analysis was adjusted for Baseline, region, sex, age, treatment, visit, visit by Baseline interaction and visit by treatment interaction. Visit 3 values were taken as Baseline value and change from Baseline was defined as the difference between the value of the endpoint at the time point of interest and the Baseline value. Statistical analysis was performed using the mixed model repeated measures (MMRM) model and least square mean and standard error were calculated. The analysis was performed on ITT Population which comprised of all participants randomized to treatment and who received at least one dose of study medication.
Time Frame: Baseline and Week 24
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Liter (L)
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 487 | 487 | 479
Liter (L) | 0.019 (0.0107) | 0.000 (0.0108) | -0.104 (0.0109)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Non-Inferiority or Equivalence — Non-inferiority was defined if the lower bound of the 95% CI for the difference between mean change from Baseline in clinic visit PM FEV1 for FF/VI and FP/S was more than -100 milliliter (mL); Least square mean change difference = 0.019, 95% CI 2-sided [-0.011 to 0.049]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, Mixed Models Analysis; Least square mean change difference = 0.123, 95% CI 2-sided [0.093 to 0.153]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, Mixed Models Analysis; Least square mean change difference = 0.104, 95% CI 2-sided [0.074 to 0.134]

2. Primary Outcome: Change From Baseline in PM FEV1 Using Per Protocol (PP) Population
Description: FEV1 was defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 (pre-bronchodilator and pre-dose) was measured at Baseline up to Week 24 at evening using spirometry. Repeated Measures analysis was adjusted for Baseline, region, sex, age, treatment, visit, visit by Baseline interaction and visit by treatment interaction. Visit 3 values were taken as Baseline value and change from Baseline was defined as the difference between the value of the endpoint at the time point of interest and the Baseline value. Statistical analysis was performed using the MMRM models and least square mean and standard error were calculated. The analysis was performed on PP Population which comprised of all participants in the ITT Population who did not had any full protocol deviations.
Time Frame: Baseline and Week 24
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 425 | 426 | 419
L | 0.020 (0.0120) | 0.014 (0.0120) | -0.099 (0.0121)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Non-Inferiority or Equivalence — Non-inferiority was defined if the lower bound of the 95% CI for the difference between mean change from Baseline in clinic visit for FF/VI and FP/S was more than -100 mL; Least square mean change difference = 0.006, 95% CI 2-sided [-0.027 to 0.040]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, Mixed Models Analysis; Least square mean change difference = 0.120, 95% CI 2-sided [0.086 to 0.153]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, Mixed Models Analysis; Least square mean change difference = 0.113, 95% CI 2-sided [0.080 to 0.147]

3. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods
Description: The number of inhalations of rescue medication used during the day and night were recorded by participants using an electronic diary (e-diary). A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week treatment period minus the Baseline value. Statistical analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of Baseline, region, sex, age and treatment and least square mean and standard error were calculated.
Time Frame: Baseline and Weeks 1-24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 500 | 498 | 496
Percentage of rescue-free 24-hr periods | -3.0 (0.62) | -4.2 (0.62) | -5.7 (0.62)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Other; Least square mean change difference = 1.2, 95% CI 2-sided [-0.5 to 3.0]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.002, ANCOVA; Least square mean change difference = 2.7, 95% CI 2-sided [0.9 to 4.4]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.106, ANCOVA; Least square mean change difference = 1.4, 95% CI 2-sided [-0.3 to 3.2]

4. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods
Description: Change from Baseline in the percentage of symptom-free 24 hour period was evaluated. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week treatment period minus the Baseline value.Statistical analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age and treatment and least square mean and standard error were calculated.
Time Frame: Baseline and Weeks 1-24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24 hour perio
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 500 | 498 | 496
Percentage of symptom-free 24 hour perio | -3.5 (0.67) | -4.7 (0.67) | -6.2 (0.67)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Other; Least square mean change difference = 1.2, 95% CI 2-sided [-0.7 to 3.1]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.004, ANCOVA; Least square mean change difference = 2.7, 95% CI 2-sided [0.8 to 4.5]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.115, ANCOVA; Least square mean change difference = 1.5, 95% CI 2-sided [-0.4 to 3.3]

5. Secondary Outcome: Change From Baseline in Morning (Ante Meridiem [AM]) Peak Expiratory Flow (PEF)
Description: PEF was measured using an electric flow meter each morning. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 24-week treatment period minus the Baseline value. Statistical analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age and treatment and least square mean and standard error were calculated.
Time Frame: Baseline and Weeks 1-24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Liter per minute (L/min)
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 501 | 499 | 497
Liter per minute (L/min) | 8.9 (1.48) | 3.7 (1.49) | -12.6 (1.49)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Other; Least square mean change difference = 5.2, 95% CI 2-sided [1.1 to 9.4]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, ANCOVA; Least square mean change difference = 21.5, 95% CI 2-sided [17.4 to 25.6]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, ANCOVA; Least square mean change difference = 16.3, 95% CI 2-sided [12.2 to 20.4]

6. Secondary Outcome: Percentage of Participants With Asthma Control Test (ACT) Score Greater Than or Equal to 20
Description: The ACT was a five-item questionnaire developed as a measure of participant's asthma control. The percentage of participants controlled, defined as having ACT score greater than or equal to 20 at the end of Week 24 were analyzed using logistic regression model with covariates of Baseline ACT score, region, sex, age and treatment group.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 471 | 467 | 461
Percentage of participants | 92 | 93 | 91
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Other; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.53 to 1.54]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.595, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.69 to 1.90]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p = 0.372, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.75 to 2.12]

7. Secondary Outcome: Change From Baseline in PM PEF
Description: PEF was measured using an electric flow meter each evening. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily PM PEF over the 24-week treatment period minus the Baseline value. Statistical analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age and treatment and least square mean and standard error were calculated.
Time Frame: Baseline and Weeks 1-24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
Number analyzed (Participants) | 501 | 498 | 496
L/min | 5.5 (1.55) | 0.5 (1.55) | -13.7 (1.55)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg Once Daily vs FP/S 250/50 mcg Twice Daily; Test type: Other; Least square mean change difference = 5.0, 95% CI 2-sided [0.7 to 9.3]
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg Once Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, ANCOVA; Least square mean change difference = 19.2, 95% CI 2-sided [14.9 to 23.5]
Statistical Analysis 3: Comparison: FP/S 250/50 mcg Twice Daily vs FP 250 mcg Twice Daily; Test type: Other; p < 0.001, ANCOVA; Least square mean change difference = 14.2, 95% CI 2-sided [9.9 to 18.5]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the follow up contact one week after completion of study medication (Up to Week 25).
Description: AEs and SAEs were collected in ITT Population
Arm/Group | FF/VI 100/25 mcg Once Daily | FP/S 250/50 mcg Twice Daily | FP 250 mcg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/504 | 0/501 | 0/499
Serious Adverse Events (participants affected / at risk) | 6/504 | 4/501 | 5/499
Other Adverse Events (participants affected / at risk) | 126/504 | 123/501 | 124/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 mcg Once Daily (N=504) | FP/S 250/50 mcg Twice Daily (N=501) | FP 250 mcg Twice Daily (N=499)
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 mcg Once Daily (N=504) | FP/S 250/50 mcg Twice Daily (N=501) | FP 250 mcg Twice Daily (N=499)
Bronchitis (Infections and infestations) | 20 | 10 | 13
Influenza (Infections and infestations) | 9 | 12 | 19
Nasopharyngitis (Infections and infestations) | 61 | 67 | 57
Pharyngitis (Infections and infestations) | 15 | 13 | 18
Headache (Nervous system disorders) | 41 | 37 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.